CLINICAL TRIAL: NCT00728546
Title: The Application of the N-acetyltransferase 2 (NAT2) Genotyping in Re-challenge Protocol of Isoniazid (INH) Titration in Patients With Anti-TB Medications-induced Hepatitis
Brief Title: NAT2 in Re-challenge of INH in Patients With Hepatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080515M
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Tuberculosis; Hepatotoxicity
Keywords: tuberculosis; isoniazid; Arylamine N-acetyl transferase; genotyping; hepatotoxicity; pharmacogenetics
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- INA dose adjustment, NAT2 (Experimental): The dose of the re-challenged INH is followed by the results of the genotyping of NAT2 in each patient.
  Interventions: Drug: Isoniazid (Rifinah)

INTERVENTIONS:
Drug: Isoniazid (Rifinah) — The dose of the re-challenged INH is followed by the results of the genotyping of NAT2 in each patient.
  Other Names: Isoniazid; Rifinah

SUMMARY:
Apply the information of NAT2 genotyping into the re-challenge protocol of INH titration in patients with anti-TB medication induced hepatitis.

DETAILED DESCRIPTION:
adjusting INH dose according to NAT2 genotyping and serum concentration of INH.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old
* Taken INH for more than 1 week
* Abnormal liver function

Exclusion criteria:

* Rule out the INH induced liver abnormality
* Existing reasons to cause liver abnormality other than TB-medication
* Taking drugs which interact with INH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Decrease the events of hepatotoxicity when patients are re-challenged with INH | 6-12 months

SECONDARY OUTCOMES:
economics evaluation of performing pharmacogenetics screening in practice | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiuan Shen, Ph.D., Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan